CLINICAL TRIAL: NCT04863430
Title: Apatinib with Oxaliplatin and S-1 Treatment for Advanced Hepatoid Adenocarcinoma of the Stomach
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The anti-PD-1 agents were proved effective by several clinical trials and recommended to treat gastric cancer. In order to protect the interest of patients, this trial was withdrawn after carefully discussion with all investigators.
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhang, Dean of VIP2 Gastrointestinal Cancer Division of Medical Department, Beijing Cancer Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC01
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; Oxaliplatin; Injections; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apatinib with chemotherapy (Experimental): Apatinib with oxaliplatin and S-1 treatment
  Interventions: Drug: Apatinib; Drug: Oxaliplatin; Drug: S1

INTERVENTIONS:
Drug: Apatinib — 500mg oral qd
  Other Names: Apatinib Mesylate Tablets
Drug: Oxaliplatin — 130mg/m^2 administered as IV infusion on Days 1 of each 21-day cycle
  Other Names: Oxaliplatin for Injection
Drug: S1 — According to body surface area,(<1.5m^2) 40mg or (≥1.5m^2)50mg bid oral on Day 1-14 of each 21-day cycle
  Other Names: Tegafur Gimeracil Oteracil Potassium Capsule

SUMMARY:
Gastric cancer is a highly heterogeneous tumor. The most commonly used clinical classifications of gastric cancer are Lauren classification (intestinal, diffuse, mixed) and World Health Organization(WHO) classification (papillary adenocarcinoma, tubular adenocarcinoma, mucinous glands cancer and low-adhesion cancer). Hepatoid adenocarcinoma of the stomach (HAS) is a special and rare type of gastric cancer.

Compared with ordinary gastric cancer, HAS has unique clinicopathological characteristics, prone to liver metastasis and lymph node metastasis, has a highly aggressive and malignant biological behavior, a worse prognosis than alpha fetoprotein(AFP) normal gastric cancer, and is easily confused with hepatocellular carcinoma(HCC). There is the possibility of misdiagnosis and mistreatment, so it has gradually attracted people's attention. Most of the domestic and foreign literature on HAS in the past 30 years are retrospective cases or small sample reports, and there are few prospective studies. There is no standard treatment plan for HAS. The main treatment is based on gastric adenocarcinoma. The clinical treatment principle is a comprehensive treatment plan with surgical resection as the mainstay, supplemented by systemic chemotherapy and local interventional therapy. This type of gastric cancer has a relatively high degree of malignancy, rapid progress of the disease, and easy recurrence after surgery. There is no standard treatment plan in China and other foreign countries.

The aim of this study was to evaluate the efficacy and safety of apatinib with oxaliplatin and S-1 treatment advanced hepatoid adenocarcinoma of the stomach.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 70 years old, no gender limitation;
2. Histopathological diagnosis of locally advanced, recurrent or metastatic HAS (pathological histomorphology and immunohistochemical diagnosis of AFP, sal-like 4(SALL4), Hep, glypican-3(GPC3), etc.);
3. Immunohistochemical(IHC) human epidermal growth factor receptor-2 (HER2) negative persons; HER2 positive is defined as IHC 3+ or IHC 2+ and fluorescence in situ hybridization(FISH)+, and FISH positive is defined as the ratio of HER2 gene copy number to chromosome 17 centromere(CEP17) signal number ≥2.0;
4. According to the RECIST 1.1 standard, at least one measurable lesion (spiral CT scan ≥10mm);
5. ECOG performance status(PS): 0-2 points;
6. The expected survival time is ≥3 months;
7. The main organs are functionally normal, without serious blood, heart, lung, liver, kidney dysfunction and immune deficiency disease. The blood test meets the following requirements; (1) Routine blood examination, which must be met (no blood transfusion within 14 days);

   1. HGB≥100g/L;
   2. WBC≥4.0×10^9/L; absolute neutrophil count(ANC) ≥2.0×10^9/L;
   3. PLT≥2.0×10^9/L; (2) The biochemical inspection must meet the following standards:

   <!-- -->

   1. BIL≤1.5 times the upper limit of normal (ULN);
   2. Alanine aminotransferase(ALT) and aspartate aminotransferase(AST)≤2.5×ULN; if there is liver metastasis, ALT and AST≤5×ULN;
   3. serum Cr≤1.5×ULN, endogenous creatinine clearance≥50ml/min (Cockcroft-Gault formula); (3) Occult blood in stool (-); (4) Urine routine is normal, or urine protein <(++), or 24-hour urine protein <1.0g;
8. The coagulation function is normal, without active bleeding and thrombosis disease;

   1. International standardized ratio INR≤1.5×ULN;
   2. Partial thromboplastin time APTT≤1.5×ULN;
   3. Prothrombin time PT≤1.5×ULN;
9. Female subjects with fertility and male subjects whose partner is a female of childbearing age who need to take effective contraceptive measures during the study treatment period and at least 6 months after the last use of the study drug;
10. Subjects voluntarily participate in this study and sign an informed consent form (ICF);
11. Those who have good compliance and can follow up as required by the plan.

Exclusion Criteria:

1. Various types of liver inflammatory diseases (especially hepatitis A, B, and C viral hepatitis active period) and other diseases that may produce AFP such as liver cirrhosis;
2. Germ cell tumors;
3. Have previously received any regimen of palliative chemotherapy for gastric cancer;
4. Have previously received apatinib treatment;
5. S-1 and/or oxaliplatin have been used in the past 6 months;
6. Those who have hypertension and cannot be reduced to the normal range after treatment with antihypertensive drugs (shrinking Pressure>140mmHg or diastolic pressure>90mmHg);
7. Suffering from coronary heart disease ≥2 grade, arrhythmia corrected QT interval(QTc) interval prolonged male> 450ms, female;>470ms) and cardiac insufficiency;
8. There are many factors that affect the absorption of oral drugs (such as inability to swallow, nausea and vomiting, chronic abdominal Diarrhea and intestinal obstruction, etc.);
9. Patients at risk of gastrointestinal bleeding or those with a history of gastrointestinal bleeding within 1 month;
10. Abnormal blood coagulation function (INR>1.5×ULN, activated partial thromboplastin time(APTT)>1.5×ULN), those with bleeding tendency;
11. Those with thrombotic diseases or receiving anticoagulant treatment;
12. Those with peripheral sensitive neuropathy with dysfunction;
13. Central nervous system metastasis;
14. Pregnant or lactating women;
15. Those who have participated in other clinical research in the past 30 days;
16. Other patients considered by the treating physician to be unsuitable for inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | Estimate up to 2 years.
  The percentage of patients having a complete response(CR) or a partial response(PR) to protocol treatment. Objective response will be measured by RECIST 1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | Estimate up to 5 years.
  The length of time from enrollment until the time of death.
Progression-free Survival (PFS) | Estimate up to 2 years.
  The time from enrollment to the first documented disease progression per RECIST 1.1 based on investigator assessment, or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | Estimate up to 2 years.
  The percentage of the participants in the analysis population who had a confirmed CR or PR or stable disease(SD) according to RECIST 1.1 based on investigator assessment.
Adverse events | Estimate up to 2 years.
  The incidence of adverse events and the incidence of severe adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital / Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No